CLINICAL TRIAL: NCT02302339
Title: A Phase 2 Study of Glembatumumab Vedotin, an Anti-gpNMB Antibody-drug Conjugate, as Monotherapy or in Combination With Immunotherapies in Patients With Advanced Melanoma
Brief Title: A Study of Glembatumumab Vedotin as Monotherapy or in Combination With Immunotherapies in Patients With Advanced Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Development of glembatumumab vedotin was discontinued
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDX011-05
Record Dates: First submitted 2014-11-19; First posted 2014-11-27 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Melanoma
Keywords: Advanced melanoma; Unresectable melanoma; Metastatic melanoma; Targeted Treatment for melanoma; GPNMB; CDX-011; Glembatumumab vedotin; Antibody-drug-conjugate; Skin neoplasm; Varlilumab; CDX-1127
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — glembatumumab vedotin; varlilumab; KPNA1 protein, human; Nivolumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Glembatumumab vedotin (Experimental): glembatumumab vedotin administered as an intravenous infusion on Day 1 of each 21 day cycle.
  Interventions: Drug: glembatumumab vedotin
- Glembatumumab vedotin and varlilumab (Experimental): glembatumumab vedotin administered as an intravenous infusion on Day 1 of each 21 day cycle. Varlilumab administered as an intravenous infusion on Day 1 of cycles 1, 2, 4, 6, 8 and 10.
  Interventions: Drug: glembatumumab vedotin and varlilumab
- Glembatumumab vedotin and PD-1 targeted checkpoint inhibitor (Experimental): glembatumumab vedotin administered as an intravenous infusion on Day 1 of each 21 day cycle. Nivolumab OR pembrolizumab administered according to institutional standard of care.
  Interventions: Drug: glembatumumab vedotin and PD-1 targeted checkpoint inhibitor (nivolumab OR pembrolizumab)
- Glembatumumab vedotin and CDX-301 (Experimental): glembatumumab vedotin administered as an intravenous infusion on Day 1 of each 21 day cycle. CDX-301 is injected once a day for five days before cycles 1 and 2.
  Interventions: Drug: glembatumumab vedotin and CDX-301

INTERVENTIONS:
Drug: glembatumumab vedotin
  Other Names: Cohort 1
  Arms: Glembatumumab vedotin
Drug: glembatumumab vedotin and varlilumab
  Other Names: Cohort 2
  Arms: Glembatumumab vedotin and varlilumab
Drug: glembatumumab vedotin and PD-1 targeted checkpoint inhibitor (nivolumab OR pembrolizumab)
  Other Names: Cohort 3
  Arms: Glembatumumab vedotin and PD-1 targeted checkpoint inhibitor
Drug: glembatumumab vedotin and CDX-301
  Other Names: Cohort 4
  Arms: Glembatumumab vedotin and CDX-301

SUMMARY:
This study will examine the effectiveness and safety of glembatumumab vedotin as monotherapy or in combination with immunotherapies in patients with advanced melanoma.

DETAILED DESCRIPTION:
Glembatumumab vedotin consists of an antibody attached to a drug, monomethyl auristatin E (MMAE), that can kill cancer cells. The fully human antibody is designed to deliver the drug to cancer cells by attaching to a protein called glycoprotein NMB (gpNMB) that is expressed on the cancer cell. The MMAE is then released inside of the cell, where it interferes with cell growth and can lead to cell death of the targeted cell, as well as neighboring cells. Varlilumab is a fully human antibody that binds to CD27. This antibody allows the body's immune system to work against cancer cells. Nivolumab is a fully human antibody and pembrolizumab is a humanized antibody. Both bind to PD-1. CDX-301 is a fully human protein that helps boost production of certain white blood cells. This protein allows the body's immune system to work against tumor cells.

Eligible patients who enroll in the study will receive treatment with one of the following: glembatumumab vedotin, glembatumumab vedotin and varlilumab, glembatumumab vedotin and CDX-301 or glembatumumab vedotin and either nivolumab OR pembrolizumab.

All patients enrolled in the study will be closely monitored to determine if their cancer is responding to treatment and for any side effects that may occur.

ELIGIBILITY:
Inclusion Criteria:

Among other criteria, patients must meet all of the following conditions to be eligible for the study:

* Unresectable, histologically-confirmed advanced (Stage III or Stage IV) melanoma
* Disease progression during or after the last anticancer therapy received. For Cohort 3, progression must have occurred during the PD-1 targeted CPI (checkpoint inhibitor) treatment and the investigator has deemed it appropriate to continue treatment with the PD-1 targeted CPI beyond confirmed disease progression
* No more than one prior chemotherapy-containing regimen for advanced disease.
* Prior treatments received must include at least one CPI inhibitor (e.g., anti-CTLA-4, PD-1-, PD-L1-targeted immunotherapy) and for patients with a BRAF mutation at least one BRAF- or MEK-targeted therapy, unless patients are not candidates for, or refused, these therapies. For cohort 3, prior treatment received must include a PD-1 targeted CPI administered during the most recent disease progression and for patients with BRAF mutation at least one BRAF- or MEK-targeted therapy when appropriate
* The study site will submit paraffin-embedded tumor tissue obtained from the patient for gpNMB analysis. Patients may require a biopsy if recent tumor tissue is not available. Patients in cohort 2 and 3 must submit a recently obtained biopsy of the skin fold for gpNMB analysis. Patients in Cohort 4 will submit a tumor tissue sample while on study.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 1
* Adequate bone marrow, liver and renal function.

Exclusion Criteria:

Among other criteria, patients who meet any of the following conditions are NOT eligible for the study:

* Previously received glembatumumab vedotin (CR011-vcMMAE, CDX-011) or other MMAE-containing agents
* Treatment with the following therapies before the planned start of study treatment:

  1. BRAF or MEK inhibitors within 2 weeks
  2. Monoclonal based therapies within 4 weeks except for the PD-1 targeted checkpoint inhibitor in cohort 3
  3. Immunotherapy (tumor vaccine, cytokine, or growth factor given to control the cancer) within 2 weeks
  4. Chemotherapy within 21 days or at least 5 half-lives (whichever is longer)
  5. Investigational therapy within 2 weeks (or at least 5 half-lives, whichever is longer)
* Patients with ocular melanoma
* Neuropathy that is moderate (Grade 2) or worse.
* Cancer that has spread to the brain or spine will be discussed with the study sponsor and may exclude patients from the trial.
* History of another cancer except:

  1. Patients with adequately treated and cured non-melanoma skin cancer or in situ cancer
  2. Patients with any other cancer from which the patient has been disease-free for ≥ 3 years
* Significant cardiovascular disease
* Previously received varlilumab or any other anti-CD27 mAb (Cohort 2 only)
* Active systemic infection requiring treatment
* Treatment with immunosuppressive medications within 4 weeks or corticosteroids within two weeks
* Patients with interstitial lung disease (Cohort 3 only)
* Patients with active diverticulitis (Cohort 3 only)
* Any non-study vaccination within 4 weeks, or influenza vaccine within 2 weeks, prior to CDX-301 dosing (Cohort 4 only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2014-11; Primary Completion 2018-06-14 (Actual); Study Completion 2018-10-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Northern California Melanoma Center/St. Mary's Medical Center, San Francisco, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Northside Hospital Cancer Institute, Atlanta, Georgia
  - University of Chicago Medicine, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - New York University School of Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Baylor Research Institute-Sammons Cancer Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Glembatumumab Vedotin: glembatumumab vedotin administered as an intravenous infusion on Day 1 of each 21 day cycle.
  glembatumumab vedotin
- Glembatumumab Vedotin and Varlilumab: glembatumumab vedotin administered as an intravenous infusion on Day 1 of each 21 day cycle. Varlilumab administered as an intravenous infusion on Day 1 of cycles 1, 2, 4, 6, 8 and 10.
  glembatumumab vedotin and varlilumab
- Glembatumumab Vedotin and PD-1 Targeted Checkpoint Inhibitor: glembatumumab vedotin administered as an intravenous infusion on Day 1 of each 21 day cycle. Nivolumab OR pembrolizumab administered according to institutional standard of care.
  glembatumumab vedotin and PD-1 targeted checkpoint inhibitor (nivolumab OR pembrolizumab)
- Glembatumumab Vedotin and CDX-301: glembatumumab vedotin administered as an intravenous infusion on Day 1 of each 21 day cycle. CDX-301 is injected once a day for five days before cycles 1 and 2.
  glembatumumab vedotin and CDX-301
Period: Overall Study
Arm/Group | Glembatumumab Vedotin | Glembatumumab Vedotin and Varlilumab | Glembatumumab Vedotin and PD-1 Targeted Checkpoint Inhibitor | Glembatumumab Vedotin and CDX-301
Started | 62 | 34 | 29 | 7
Completed | 61 | 32 | 28 | 7
Not Completed | 1 | 2 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glembatumumab Vedotin | Glembatumumab Vedotin and Varlilumab | Glembatumumab Vedotin and PD-1 Targeted Checkpoint Inhibitor | Glembatumumab Vedotin and CDX-301 | Total
Number analyzed (Participants) | 62 | 34 | 29 | 7 | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 26 | 21 | 11 | 6 | 64
  >=65 years | 36 | 13 | 18 | 1 | 68
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 14 | 11 | 4 | 57
  Male | 34 | 20 | 18 | 3 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 2 | 0 | 9
  Not Hispanic or Latino | 57 | 32 | 27 | 7 | 123
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 61 | 32 | 27 | 6 | 126
  Black or African American | 1 | 0 | 0 | 1 | 2
  Asian | 0 | 1 | 0 | 0 | 1
  Other | 0 | 1 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of patients who achieved best overall response of complete or partial response. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST version 1.1), Complete Response (CR) = disappearance of all target lesions and non-target lesions, Partial Response (PR), >= 30% decrease in the sum of the longest diameter of target lesions with no progression in non-target lesions and no new lesions. ORR was the primary outcome for Cohorts 1-3 and a secondary outcome for Cohort 4.
Time Frame: Every 6 to 9 weeks following treatment initiation until disease progression.
Population: Response evaluable (at least one dose and a post treatment disease assessment)
Measure: Count of Participants; unit: Participants
Arm/Group | Glembatumumab Vedotin | Glembatumumab Vedotin and Varlilumab | Glembatumumab Vedotin and PD-1 Targeted Checkpoint Inhibitor | Glembatumumab Vedotin and CDX-301
Number analyzed (Participants) | 62 | 31 | 28 | 5
Participants | 7 | 1 | 4 | 0

2. Primary Outcome: Adverse Events of the Combination of Glembatumumab Vedotin and CDX-301 (in Cohort 4).
Description: The percentage of patients experiencing one or more adverse events.
Time Frame: Up to 18 months following the screening visit
Measure: Count of Participants; unit: Participants
Arm/Group | Glembatumumab Vedotin and CDX-301
Number analyzed (Participants) | 7
Participants
  Leukopenia | 1
  Abdominal pain | 1
  Constipation | 2
  Dyspepsia | 2
  Nausea | 1
  Stomatitis | 1
  Vomiting | 1
  Fatigue | 3
  Hepatic pain | 1
  Mucosal infection | 1
  Urinary tract infection | 1
  Alanine aminotransferase increased | 2
  Aspartate aminotransferase increased | 3
  Blood alkaline phosphatase increased | 1
  Neutrophil count decreased | 1
  Platelet count decreased | 1
  Weight decreased | 1
  Decreased appetite | 1
  Hyperglycemia | 1
  Hyperuricemia | 1
  Hypokalemia | 1
  Myalgia | 1
  Pain in extremity | 1
  Peripheral sensory neuropathy | 1
  Anxiety | 1
  Depression | 1
  Vaginal hemorrhage | 1
  Vulvovaginal pain | 1
  Epistaxis | 1
  Alopecia | 3
  Rash erythematous | 1
  Rash maculopapular | 3
  Skin discoloration | 1
  Hypertension | 1

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR is the number of months from the time criteria are first met for either CR or PR, until the first date that PD is objectively documented per RECIST 1.1.
Time Frame: From start date of partial or complete response (whichever is achieved first) to first date that recurrent of progressive disease is objectively documented, assessed up to 18 months.
Population: Number of patients analyzed are the number of patients who achieved an objective response per Cohort. The response was observed at the last measurement without further follow up due to study closure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Glembatumumab Vedotin | Glembatumumab Vedotin and Varlilumab | Glembatumumab Vedotin and PD-1 Targeted Checkpoint Inhibitor | Glembatumumab Vedotin and CDX-301
Number analyzed (Participants) | 7 | 1 | 4 | 0
months | 6.0 [4.1 to 27.5] | 2.2 [NA to NA] — With only 1 response achieved, it is not possible to calculate confidence intervals. | 6.2 [3.1 to 6.2] |

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from randomization to the earlier of disease progression or death due to any cause. Disease progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or progression in a non-target lesion, or the appearance of new lesions.
Time Frame: Evaluated every 6 to 9 weeks following treatment initiation until progression.
Population: Response evaluable (at least one dose and a post treatment disease assessment). The analysis was not completed for the glembatumumab + CDX-301 cohort because sufficient data were not collected to perform the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Glembatumumab Vedotin | Glembatumumab Vedotin and Varlilumab | Glembatumumab Vedotin and PD-1 Targeted Checkpoint Inhibitor | Glembatumumab Vedotin and CDX-301
Number analyzed (Participants) | 62 | 31 | 28 | 0
months | 4.4 [2.6 to 5.4] | 2.6 [1.4 to 2.9] | 4.1 [2.7 to 6.9] |

5. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is defined as the number of months from randomization to the date of death due to any cause.
Time Frame: During treatment and every 3 months from end of treatment through death or end of study
Population: Response evaluable (at least one dose and a post treatment disease assessment). The analysis was not completed for the glembatumumab + CDX-301 cohort or the glembatumumab vedotin and PD-1 targeted checkpoint inhibitor cohort because sufficient data were not collected to perform the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Glembatumumab Vedotin | Glembatumumab Vedotin and Varlilumab | Glembatumumab Vedotin and PD-1 Targeted Checkpoint Inhibitor | Glembatumumab Vedotin and CDX-301
Number analyzed (Participants) | 62 | 31 | 0 | 0
months | 8.8 [5.9 to 11.7] | 6.6 [3.2 to 8.6] |  |

6. Secondary Outcome: Correlation of Activity to gpNMB Expression
Description: To investigate if the anti-cancer activity of glembatumumab vedotin as monotherapy or in combination with immunotherapies in advanced melanoma is dependent upon the degree of gpNMB expression in tumor tissue.
Time Frame: Up to 18 months following the screening visit
Population: Analysis not completed. gpNMB expression in tumor tissue was not done.
Arm/Group | Glembatumumab Vedotin | Glembatumumab Vedotin and Varlilumab | Glembatumumab Vedotin and PD-1 Targeted Checkpoint Inhibitor | Glembatumumab Vedotin and CDX-301
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Adverse Events
Description: The percentage of patients experiencing one or more AEs will be summarized by relationship to study drug and severity.
Time Frame: Following at least one dose of study treatment through 28 days after last dose of glembatumumab vedotin, or 70 calendar days after last administration of varlilumab, CDX-301 or PD-1 targeted checkpoint inhibitor (whichever occurs latest)
Measure: Count of Participants; unit: Participants
Arm/Group | Glembatumumab Vedotin | Glembatumumab Vedotin and Varlilumab | Glembatumumab Vedotin and PD-1 Targeted Checkpoint Inhibitor | Glembatumumab Vedotin and CDX-301
Number analyzed (Participants) | 62 | 34 | 29 | 7
Participants | 61 | 34 | 29 | 7

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded from the time the patient has taken at least one dose of study treatment through (whichever occurs first) either: a) 28 - 70 calendar days after the last administration of study drug depending on the cohort; or b) initiation of alternate anticancer therapy.
Arm/Group | Glembatumumab Vedotin | Glembatumumab Vedotin and Varlilumab | Glembatumumab Vedotin and PD-1 Targeted Checkpoint Inhibitor | Glembatumumab Vedotin and CDX-301
All-Cause Mortality (participants affected / at risk) | 53/62 | 26/34 | 8/29 | 1/7
Serious Adverse Events (participants affected / at risk) | 19/62 | 14/34 | 14/29 | 2/7
Other Adverse Events (participants affected / at risk) | 61/62 | 34/34 | 29/29 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Glembatumumab Vedotin (N=62) | Glembatumumab Vedotin and Varlilumab (N=34) | Glembatumumab Vedotin and PD-1 Targeted Checkpoint Inhibitor (N=29) | Glembatumumab Vedotin and CDX-301 (N=7)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 1 | 0
Acute Coronary Syndrome (Cardiac disorders) | 0 | 0 | 1 | 0
Angina Pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0
Infusion Site Extravasation (General disorders) | 1 | 0 | 0 | 0
Multiple Organ Dysfunction Syndrome (General disorders) | 0 | 0 | 2 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 0
Hepatic Failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Atypical Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 2 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 4 | 0
Septic Shock (Infections and infestations) | 1 | 2 | 0 | 0
Skin Infection (Infections and infestations) | 1 | 0 | 0 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Neutrophil Count Decreased (Investigations) | 1 | 0 | 0 | 1
White Blood Cell Count Decreased (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 1 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0 | 1 | 0
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Intensive Care Unit Acquired Weakness (Nervous system disorders) | 0 | 1 | 0 | 0
Confusional State (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 2 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rash Macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Toxic Epidermal Necrolysis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Embolism (Vascular disorders) | 1 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Glembatumumab Vedotin (N=62) | Glembatumumab Vedotin and Varlilumab (N=34) | Glembatumumab Vedotin and PD-1 Targeted Checkpoint Inhibitor (N=29) | Glembatumumab Vedotin and CDX-301 (N=7)
Anemia (Blood and lymphatic system disorders) | 15 | 13 | 4 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 7 | 4 | 7 | 0
Atrial Fibrilation (Cardiac disorders) | 0 | 0 | 2 | 0
Palpitations (Cardiac disorders) | 4 | 0 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 2 | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 2 | 0
Vision Blurred (Eye disorders) | 3 | 1 | 2 | 0
Abdominal Distension (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 11 | 6 | 7 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 14 | 13 | 11 | 2
Diarrhoea (Gastrointestinal disorders) | 19 | 15 | 14 | 0
Dry Mouth (Gastrointestinal disorders) | 6 | 1 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 3 | 3 | 2
Flatulence (Gastrointestinal disorders) | 1 | 2 | 2 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 4 | 1 | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 23 | 12 | 16 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Stomatits (Gastrointestinal disorders) | 7 | 2 | 6 | 1
Vomiting (Gastrointestinal disorders) | 12 | 10 | 8 | 1
Asthenia (General disorders) | 4 | 2 | 2 | 0
Chills (General disorders) | 3 | 2 | 7 | 0
Fatigue (General disorders) | 26 | 22 | 11 | 3
Influenza Like Illness (General disorders) | 3 | 2 | 0 | 0
Malaise (General disorders) | 0 | 0 | 2 | 0
Non-Cardiac Chest pain (General disorders) | 2 | 2 | 2 | 0
Oedema Peripheral (General disorders) | 9 | 3 | 3 | 0
Pain (General disorders) | 4 | 4 | 1 | 0
Pyrexia (General disorders) | 6 | 7 | 6 | 0
Hepatic Pain (Hepatobiliary disorders) | 1 | 1 | 1 | 1
Candida Infection (Infections and infestations) | 2 | 2 | 4 | 0
Eye Infection (Infections and infestations) | 0 | 0 | 2 | 0
Mucosal Infection (Infections and infestations) | 0 | 0 | 1 | 1
Oral Candidiasis (Infections and infestations) | 2 | 6 | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 2 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 3 | 2 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 0
Procedural Site Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 3 | 5 | 6 | 2
Aspartate Aminotransferase Increased (Investigations) | 8 | 4 | 7 | 3
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 2 | 1 | 1
Blood Creatinine Increased (Investigations) | 5 | 0 | 1 | 0
Lymphocyte Count Decreased (Investigations) | 4 | 1 | 1 | 0
Neutrophil Count Decreased (Investigations) | 14 | 5 | 8 | 1
Platelet Count Decreased (Investigations) | 1 | 0 | 1 | 1
Weight Decreased (Investigations) | 10 | 6 | 7 | 1
White Blood Cell Count Decreased (Investigations) | 8 | 4 | 7 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 23 | 13 | 11 | 1
Dehydration (Metabolism and nutrition disorders) | 9 | 7 | 6 | 0
Hyperglaecemia (Metabolism and nutrition disorders) | 5 | 4 | 3 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 1 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 | 1 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 1 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 3 | 3 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 1 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 11 | 5 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 0 | 3 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 4 | 8 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 1 | 3 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Muscle Spasma (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 8 | 0 | 3 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 0
Muskuloskeletal Pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 3 | 4 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 | 2 | 7 | 1
Carpal Tunnel Syndrome (Nervous system disorders) | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 6 | 2 | 3 | 0
Dysgeusia (Nervous system disorders) | 6 | 2 | 7 | 0
Encephalopathy (Nervous system disorders) | 0 | 2 | 2 | 0
Headache (Nervous system disorders) | 9 | 5 | 5 | 0
Paraesthesia (Nervous system disorders) | 4 | 1 | 2 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 27 | 8 | 10 | 1
Seizure (Nervous system disorders) | 0 | 2 | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 2 | 5 | 1
Confusional State (Psychiatric disorders) | 1 | 4 | 1 | 0
Depression (Psychiatric disorders) | 3 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 11 | 3 | 7 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 2 | 0
Acute Kidney Injury (Renal and urinary disorders) | 3 | 3 | 1 | 0
Micronutrition Urgency (Renal and urinary disorders) | 0 | 0 | 2 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 2 | 0 | 0
Vaginal Hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vuvlovaginal Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 3 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 5 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 5 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 30 | 15 | 15 | 3
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 5 | 2 | 1 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 15 | 10 | 13 | 0
Pruritis Generalised (Skin and subcutaneous tissue disorders) | 2 | 8 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 9 | 4 | 4 | 0
Rash Erythaemous (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 1
Rash Generalised (Skin and subcutaneous tissue disorders) | 6 | 3 | 6 | 0
Rash Mascular (Skin and subcutaneous tissue disorders) | 4 | 1 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 11 | 13 | 11 | 3
Rash Pruritic (Skin and subcutaneous tissue disorders) | 3 | 2 | 1 | 0
Skin Discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 3 | 0 | 2 | 0
Hypertension (Vascular disorders) | 2 | 1 | 0 | 1
Hypotension (Vascular disorders) | 7 | 1 | 2 | 0

LIMITATIONS AND CAVEATS:
Study was discontinued early, leading to small number of subjects analyzed in Cohort 4 and minimal patient follow up in Cohorts 3 and 4.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-28): https://cdn.clinicaltrials.gov/large-docs/39/NCT02302339/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/39/NCT02302339/SAP_001.pdf